CLINICAL TRIAL: NCT06039631
Title: Neoadjuvant Immunotherapy And Chemotherapy Followed By Concurrent Chemoradiation Or Organ Preservation Surgery In Locally Advanced Laryngeal Cancer And Hypopharyngeal Cancer
Brief Title: Neoadjuvant Chemoimmunotherapy Followed By Radiation Or Organ Preservation Surgery In Laryngeal/Hypopharyngeal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Fudan University Eye Ear Nose and Throat Hospital (Unknown); Shanghai Zhongshan Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Ruijin Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yu Wang, M.D., Chair, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Larynx-IO 2.0
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Larynx Cancer; Hypopharyngeal Cancer
Keywords: organ preservation; PD-1 inhibitor; Immunotherapy; Neoadjuvant chemotherapy; Induction chemotherapy; larynx presrvation surgery
MeSH Terms: conditions — Laryngeal Neoplasms; Hypopharyngeal Neoplasms | interventions — Surgical Procedures, Operative; Radiation; toripalimab

STUDY DESIGN:
Intervention Model Description: the selection trial design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Organ preservation surgery (Experimental): In the surgical group, patients will undergo curative surgery for laryngeal/hypopharyngeal cancer along with cervical lymph node dissection. Organ preservation surgery is recommended, and the specific surgical approach will be chosen based on individual case characteristics and the treatment protocols followed at our center. Depending on postoperative pathology results, adjuvant radiotherapy or concurrent radiochemotherapy may be administered as deemed necessary. If postoperative pathology indicates extracapsular invasion of lymph nodes or positive surgical margins, concurrent radiochemotherapy based on cisplatin is recommended. Starting three weeks after the completion of radiotherapy, patients will receive adjuvant immunotherapy using a specific protocol of toripalimab at a dose of 240 mg every 3 weeks for a total of 8 cycles.
  Interventions: Procedure: Surgery; Radiation: Radiation; Drug: Toripalimab
- Concurrent chemoradiation (Other): In the concurrent radiochemotherapy group, patients will undergo target delineation based on the scope before induction chemotherapy. Radiotherapy will be administered at a total dose of 70 Gy over 35 fractions, and concurrent chemotherapy will involve weekly administration of cisplatin. Starting three weeks after the completion of radiotherapy, patients will receive adjuvant immunotherapy using a specific protocol of toripalimab at a dose of 240 mg every 3 weeks for a total of 8 cycles.
  Interventions: Radiation: Radiation; Drug: Toripalimab

INTERVENTIONS:
Procedure: Surgery — In the surgical group, patients will undergo curative surgery for laryngeal/hypopharyngeal cancer along with cervical lymph node dissection. Organ preservation surgery is recommended.
  Arms: Organ preservation surgery
Radiation: Radiation — In the surgical group, depending on postoperative pathology results, adjuvant radiotherapy or concurrent radiochemotherapy may be administered as deemed necessary. If postoperative pathology indicates extracapsular invasion of lymph nodes or positive surgical margins, concurrent radiochemotherapy based on cisplatin is recommended.
  In the concurrent radiochemotherapy group, patients will undergo target delineation based on the scope before induction chemotherapy. Radiotherapy will be administered at a total dose of 70 Gy over 35 fractions, and concurrent chemotherapy will involve weekly administration of cisplatin at a dosage of 30 mg/m².
Drug: Toripalimab — In the both groups, starting three weeks after the completion of radiotherapy, patients will receive adjuvant immunotherapy using a specific protocol of toripalimab at a dose of 240 mg every 3 weeks for a total of 8 cycles.

SUMMARY:
In the global landscape of cancer, head and neck malignancies are highly prevalent, with 878,000 new cases and 444,000 deaths recorded in 2020. Notably, laryngeal and hypopharyngeal cancers contribute to around 30% of these instances. More than 50% of patients are diagnosed with locally advanced disease, necessitating intensive treatments that significantly impact their quality of life. Despite these efforts, the prognosis for laryngeal and hypopharyngeal cancers remains grim, with a 5-year survival rate of 30% to 50%.

Past approaches focused on preserving laryngeal function and patient well-being, including minimally invasive surgery, advanced radiotherapy, and induction chemotherapy. Our prior research highlighted the effectiveness of combining toripalimab-based induction therapy and chemotherapy, followed by concurrent chemoradiotherapy or surgery. Positive short-term outcomes and manageable side effects were observed, with encouraging larynx preservation rates after one year.

Against this backdrop, the current study aims to explore neoadjuvant immunotherapy combined with chemotherapy for patients with locally advanced laryngeal and hypopharyngeal cancer. It seeks to compare the therapeutic efficacy and quality of life impacts of concurrent radiochemotherapy and organ-preserving surgery. The ultimate goal is to identify optimal strategies for future interventions.

DETAILED DESCRIPTION:
Head and neck cancer stands as one of the most prevalent forms of malignancy on a global scale. Among these, head and neck squamous cell carcinoma (HNSCC) takes precedence as the predominant histological subtype, encompassing around 90% of the total caseload. Notably, laryngeal and hypopharyngeal cancer contribute to approximately 30% of these instances. Upon initial diagnosis, a striking majority-over 50% of patients find themselves grappling with locally advanced disease, necessitating an assertive therapeutic approach that significantly impacts their overall quality of life. Despite the rigor of these treatments, the prognosis for laryngeal and hypopharyngeal cancer remains discouraging, characterized by a 5-year overall survival rate ranging between 30% and 50%.

Past endeavors have been dedicated to preserving laryngeal function and enhancing the well-being of patients, spanning from the adoption of minimally invasive and organ-conserving surgical techniques to advancements in radiotherapy and the advent of induction chemotherapy. Recent strides in immunotherapy, particularly the integration of programmed cell death protein-1 (PD-1) inhibitors, have brought about a remarkable paradigm shift in how recurrent/metastatic HNSCC is managed. Our previous investigation underscored the efficacy of the strategy involving the combination of toripalimab-based induction therapy and chemotherapy, followed by concurrent chemoradiotherapy or surgical intervention, showcasing favorable short-term outcomes and manageable adverse effects. The data further revealed highly promising larynx preservation rates at the one-year mark.

Given this backdrop, the present study seeks to delve into patients experiencing partial relief through neoadjuvant immunotherapy combined with chemotherapy in cases of locally advanced laryngeal and hypopharyngeal cancer. The study aims to compare the therapeutic efficacy and discrepancies in quality of life resulting from concurrent radiochemotherapy and organ-preserving surgical treatment. The overarching goal is to delineate optimal strategies for subsequent interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Signing of the informed consent form and willingness to comply with the study protocol.
2. Age ≥18 and ≤75 years.
3. Histologically confirmed laryngeal or hypopharyngeal squamous cell carcinoma.
4. Locally advanced laryngeal/hypopharyngeal cancer patients eligible for surgical resection (AJCC 8th edition stage: T2N+M0, T3-T4aN0-3M0).
5. Presence of at least one measurable lesion before treatment, in accordance with RECIST 1.1 criteria for "measurable lesions."
6. Patients who have received neoadjuvant immunotherapy combined with chemotherapy and have achieved a partial response (PR) in the primary lesion according to RECIST 1.1 criteria and are suitable candidates for organ preservation surgery.
7. Expected survival of more than 3 months.
8. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
9. Good organ function, meeting the following criteria:

   1. Absolute neutrophil count (ANC) ≥1.5×10^9/L.
   2. Platelet count ≥100×10^9/L.
   3. Hemoglobin ≥9 g/dL.
   4. Serum albumin ≥2.8 g/dL.
   5. Total bilirubin ≤1.5× upper limit of normal (ULN), ALT, AST, and/or ALP ≤3× ULN.
   6. Serum creatinine ≤1.5× ULN and creatinine clearance ≥60 mL/min (Cockcroft-Gault formula, see Appendix III).
   7. Activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤1.5× ULN (patients on stable doses of anticoagulation with agents like low molecular weight heparin or warfarin, and INR within the expected therapeutic range, may be included).
10. Patients with hepatitis B virus (HBV) infection, inactive/asymptomatic HBV carriers, or patients with chronic or active HBV infection with HBV DNA <500 IU/mL (or 2500 copies/mL) at screening will be allowed to participate. Patients positive for hepatitis C antibodies, if HCV-RNA is negative at screening, will be allowed to participate.
11. Females of childbearing potential must have a negative pregnancy test result in urine or serum ≤7 days before treatment initiation. They must use a medically accepted contraceptive measure (such as intrauterine device, oral contraceptives, or condoms) during the study treatment period, for at least 3 months after the last dose of toripalimab, and for at least 6 months after the last dose of chemotherapy.
12. Non-sterilized male participants must be willing to use a medically accepted contraceptive measure (such as intrauterine device, oral contraceptives, or condoms) during the study treatment period, for at least 3 months after the last dose of toripalimab, and for at least 6 months after the last dose of chemotherapy.

Exclusion Criteria:

1. History of allergic reactions to any components of toripalimab, paclitaxel, or cisplatin.
2. Pre-existing tracheostomy due to laryngeal dysfunction before treatment.
3. History of or concurrent presence of other malignancies (except for those cured and with no cancer-related survival exceeding 5 years, such as basal cell carcinoma of the skin, cervical carcinoma in situ, and papillary thyroid cancer). Patients with concurrent hypopharyngeal and esophageal cancers, where the lesions are not anatomically adjacent, will be diagnosed as having dual primary tumors and will not be eligible for inclusion.
4. Uncontrolled clinical cardiac symptoms or diseases, including:

   1. NYHA Class II or higher heart failure.
   2. Unstable angina.
   3. Myocardial infarction within the past year.
   4. Clinically significant ventricular or supraventricular arrhythmias requiring clinical intervention.
5. Previous treatment with any of the following:

   1. Use of any investigational drug within 4 weeks prior to the first dose of study treatment.
   2. Concurrent participation in another clinical trial, unless it is an observational (non-interventional) clinical trial.
   3. Requiring systemic treatment with corticosteroids (daily dose >10 mg prednisone equivalent) or other immunosuppressive medications within 2 weeks prior to the first dose of study treatment, excluding corticosteroids for localized inflammation or prophylaxis against allergies or nausea/vomiting. Other specific circumstances should be discussed with the investigator. In the absence of active autoimmune disease, inhaled or topical steroids and adrenal replacement therapy with a dose of >10 mg/day prednisone or equivalent are allowed.
   4. Vaccination with anti-tumor vaccines or administration of live vaccines within 4 weeks prior to the first dose of study treatment (for patients who received COVID-19 vaccine, a 2-week interval is required).
   5. Major surgery within 4 weeks before the first dose of study treatment or presence of severe trauma.
6. Failure to recover to ≤ Grade 1 toxicity per CTCAE (except for alopecia and residual neuropathy related to prior platinum therapy) from previous cancer therapy or from any other cause unrelated to study/enrollment criteria.
7. Experience of severe infections (CTCAE > Grade 2) within 4 weeks before the first dose of study treatment, such as severe pneumonia requiring hospitalization, sepsis, or complicated infections. Baseline chest imaging indicating active pulmonary inflammation, presence of symptoms and signs of infection within 4 weeks before the first dose of study treatment, or requirement for oral or intravenous antibiotics to treat infection are exclusion criteria.
8. Active autoimmune disease or history of autoimmune disease, such as interstitial lung disease, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but not limited to these diseases or syndromes. However, stable dose of thyroid replacement therapy for autoimmune-mediated hypothyroidism is allowed. Stable dose of insulin for type I diabetes is allowed. Patients with vitiligo or childhood-onset asthma/allergies requiring no intervention as adults are allowed.
9. History of immune deficiency, including HIV positive test results, other acquired or congenital immunodeficiency diseases, or history of organ transplantation or allogeneic bone marrow transplantation.
10. History of interstitial lung disease (excluding radiation pneumonitis not treated with steroids), non-infectious pneumonitis.
11. Active tuberculosis infection found through medical history or CT scan, or presence of active tuberculosis infection within the past year prior to enrollment, or history of active tuberculosis infection more than 1 year ago but not formally treated.
12. Presence of active hepatitis B (HBV DNA ≥500 IU/mL or 2500 copies/mL) or hepatitis C (HCV-RNA positive with HCV-RNA levels above the lower limit of detection of the assay) infection＊.
13. Known history of substance abuse, alcohol abuse, or drug addiction.
14. Pregnant or breastfeeding women.
15. Other factors, as judged by the investigator, that may interfere with the participant's ability to comply with the study requirements or that may jeopardize the safety of the participant or the quality of the study data, including the presence of other severe diseases (including mental illness) requiring concurrent treatment, severe abnormal laboratory values, family or social factors, which might affect participant safety or data collection.

    * For participants who are HBsAg-positive and either HBV DNA-negative or with HBV DNA <500 IU/mL or 2500 copies/mL, after receiving stable antiviral treatment, they may be included in this trial (treatment should be ongoing for >2 weeks before enrollment, and continued for 6 months after the last dose of study treatment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | At two year post-randomization
  Progression-free survival is defined as the time interval from the commencement of randomization until the first documented occurrence of objective tumor progression or death due to any cause, whichever comes first.

SECONDARY OUTCOMES:
Larynx Preservation rate | At two year post-randomization
  Larynx-preservation is considered to have failed on the date of total laryngectomy, or evidence of local recurrence on primary site.
Overall Survival rate | At two year post-randomization
  Overall survival is measured as the time from the initiation of randomization to the occurrence of death due to any cause.
Quality of life | From enrollment to two year post-randomization
  Evaluated by MD Anderson Dysphagia Inventory, Voice Handicap Index 10
Adverse events | From enrollment to two year post-randomization
  Adverse events evaluated by CTCAE 5.0 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The sharing of inviduual participant data will be decided after the pubilcation of this research and the approvement of IRB of Fudan Univerisity Shanghai Cancer Center
Supporting Information: Study Protocol
Time Frame: After the pubilcation of this study and the approvement of IRB, till two years after pubilcation.
Access Criteria: The data will be assessed via contact with principal investigator.